CLINICAL TRIAL: NCT01143272
Title: Saccharomyces Boulardii for the Prevention of Antibiotic-associated Diarrhoea - Randomised, Double-blind, Placebo-controlled Trial
Brief Title: Probiotic Saccharomyces Boulardii for the Prevention of Antibiotic-associated Diarrhoea
Acronym: SacBo
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Masked independent interim analysis: completion of the trial was unlikely.
Sponsor: Bernhard Nocht Institute for Tropical Medicine (Other Government)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Stephan Ehrhardt, Lead investigator, Bernhard Nocht Institute for Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BNI-2009-01; 2009-017374-20 (EudraCT Number); ISRCTN01005546 (Registry Identifier: ISRCTN, http://www.controlled-trials.com/ISRCTN01005546); DRKS00000084 (Registry Identifier: Deutsches Register Klinischer Studien)
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Results first posted 2016-07-18 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-06

CONDITIONS: Antibiotic-associated Diarrhea; Clostridium Difficile; Diarrhea
Keywords: antibiotic; associated; diarrhoea; saccharomyces boulardii; Antibiotic-associated diarrhoea (AAD); Clostridium difficile-associated-diarrhoea (CDAD)
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saccharomyces boulardii (Active Comparator): Participants received Saccharomyces boulardii 250 mg capsules twice per day within 24 hours of initiating antibiotic treatment and continued treatment for 7 days after antibiotic discontinuation
  Interventions: Drug: Saccharomyces boulardii
- Microcristallin cellulose (Placebo Comparator): Participants received matching placebo twice per day within 24 hours of initiating antibiotic treatment and continued treatment for 7 days after antibiotic discontinuation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Saccharomyces boulardii — Units: 500 mg per day Route of administration : Oral Use Hard-Capsule
  Other Names: Perenterol® Forte
  Arms: Saccharomyces boulardii
Drug: Placebo — Placebo
  Other Names: Microcristallin cellulose; Matching capsules containing no active ingredients
  Arms: Microcristallin cellulose

SUMMARY:
When patients in hospitals receive antibiotics they often develop diarrhoea. The consequences may be grave for the patient. Thus far, no preventive measure is available. The investigators hypothesize that the apathogenic yeast Saccharomyces boulardii, administered in addition to the antibiotic, may prevent episodes of diarrhoea or may lead to less pronounced diarrhoea. To test this hypothesis, the investigators are carrying out a clinical trial in 1520 adult patients in several hospitals.

DETAILED DESCRIPTION:
Antibiotic-associated diarrhoea (AAD) is a frequent condition in hospitalised patients receiving antibiotic treatment. The same is true for Clostridium difficile-associated diarrhoea (CDAD) with even more grave consequences of increased morbidity and mortality. The development and evaluation of preventive strategies is one key public health challenge. In the absence of clinically evaluated alternatives, probiotics have been suggested to be beneficial for the prevention of AAD and CDAD. However, data have so far been inconclusive and recently published meta-analyses strongly recommended large state-of-the-art clinical trials on probiotic substances for the prevention of AAD and CDAD. Since the efficacy, side-effects and modes of action of different probiotic bacteria and yeast are strain specific, benefits and risks cannot be generalised. The non-pathogenic yeast Saccharomyces cerevisiae var. boulardii (Sac. boulardii) is considered the most promising probiotic substance for the prevention of AAD and CDAD. We carry out a randomised, placebo controlled, double blind multicentre clinical trial to evaluate Sac. boulardii for the indication of prevention of AAD and CDAD in 1520 adult, hospitalised patients.

ELIGIBILITY:
Inclusion Criteria:

* adult patient (≥ 18 years)
* patient hospitalized
* patient receives systemic antibiotic treatment
* patient contractually capable
* patient able to follow study procedures
* informed consent of patient

Exclusion Criteria:

* allergy against yeast and/or Perenterol® forte und/oder placebos containing Saccharomyces cerevisiae HANSEN CBS 5926, lactose-monohydrate, magnesium stearate, gelatine, sodium dodecyl sulfate, titan dioxide, microcrystalline cellulose.
* central venous catheter
* immunosuppression
* diarrhoea and/or chronic diarrhoea
* regular intake of Perenterol®, Perenterol® forte oder Yomogi® in the last seven days before the start of the study
* systemic antimycotic treatment
* systemic antibiotic treatment within the last 6 weeks
* no protection against conception, pregnancy, or lactation
* simultaneous participation in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 477 (Actual)
Dates: Start 2010-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Ehrhardt, MD, MPH, Principal Investigator — Bernhard Nocht Institute for Tropical Medicine, Hamburg, Germany
Locations (14):
- Germany (14):
  - Abteilung Innere Medizin, Bundeswehrkrankenhaus Ulm, Ulm, Baden-Würtemberg
  - Klinikum Bremen Ost, Klinik für Innere Medizin, Bremen, City state Bremen
  - I. Medizinische Klinik und Poliklinik, Universitätsklinikum Hamburg-Eppendorf, Hamburg, Hamburg
  - Agaplesion Diakonieklinikum Hamburg, Klinik für Innere Medizin, Hamburg, Hamburg
  - Bethesda Krankenhaus Bergedorf, Klinik für Innere Medizin, Hamburg, Hamburg
  - Diakoniekrankenhaus Rotenburg (Wümme) gGmbH, Zentrum für Pneumologie, Rotenburg (Wümme), Lower Saxony
  - Klinik und Poliklinik für Innere Medizin, Abteilung für Tropenmedizin und Infektionskrankheiten, Universitätsklinikum Rostock, Rostock, Mecklenburg-Vorpommern
  - Knappschaftskrankenhaus Bottrop, Medizinische Klinik, Bottrop, North Rhine-Westphalia
  - Abteilung Akut-Geriatrie, Ev. Krankenhaus Bethanien Iserlohn, Iserlohn, North Rhine-Westphalia
  - Klinikum Vest GmbH, Behandlungszentrum Paracelsus-Klinik Marl, Marl, North Rhine-Westphalia
  - I. Medizinische Klinik und Poliklinik, Johannes-Gutenberg-Universität Mainz, Mainz, Rhineland-Palatinate
  - Klinikum Saarbrücken, Saarbrücken, Saarland
  - Klinikum St.Georg, Klinik für Infektiologie, Tropenmedizin und Nephrologie, Leipzig, Saxony
  - Abt. Innere Medizin, Krankenhaus Reinbek, St. Adolf -Stift, Reinbek, Schleswig-Holstein

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ehrhardt S, Guo N, Hinz R, Schoppen S, May J, Reiser M, Schroeder MP, Schmiedel S, Keuchel M, Reisinger EC, Langeheinecke A, de Weerth A, Schuchmann M, Schaberg T, Ligges S, Eveslage M, Hagen RM, Burchard GD, Lohse AW. Saccharomyces boulardii to Prevent Antibiotic-Associated Diarrhea: A Randomized, Double-Masked, Placebo-Controlled Trial. Open Forum Infect Dis. 2016 Jan 29;3(1):ofw011. doi: 10.1093/ofid/ofw011. eCollection 2016 Jan. PMID 26973849
- See also: Sponsor website — http://www.bni-hamburg.de

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Saccharomyces Boulardii | Microcristallin Cellulose
Started | 246 | 231
Completed | 246 | 231
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saccharomyces Boulardii | Microcristallin Cellulose | Total
Number analyzed (Participants) | 246 | 231 | 477
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (16.5) | 56.5 (17.8) | 58.4 (17.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 102 | 208
  Male | 140 | 129 | 269
Region of Enrollment [Number; unit: participants]
  Germany | 246 | 231 | 477
Body height [Mean (Standard Deviation); unit: cm] | 171.8 (9.4) | 171.7 (10.0) | 171.7 (9.7)
Body weight [Mean (Standard Deviation); unit: kg] | 83.1 (17.0) | 83.0 (18.1) | 83.0 (17.5)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 28.1 (5.2) | 28.1 (5.6) | 28.1 (5.4)
C-reactive protein (CRP) [Mean (Standard Deviation); unit: mg/L] | 71.0 (89.3) | 72.2 (98.9) | 71.6 (93.9)
Leukocyte count [Mean (Standard Deviation); unit: 10^9 cells/L] | 10.3 (4.6) | 11.4 (6.7) | 10.8 (5.7)

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Antibiotic-associated Diarrhea Episodes
Time Frame: 29 months
Measure: Number; unit: Episodes
Arm/Group | Saccharomyces Boulardii | Microcristallin Cellulose
Number analyzed (Participants) | 246 | 231
Episodes | 21 | 19
Statistical Analysis 1: Comparison: Saccharomyces Boulardii vs Microcristallin Cellulose; Test type: Superiority or Other; p = 0.94, Regression, Cox; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.55 to 1.90]
Statistical Analysis 2: Comparison: Saccharomyces Boulardii vs Microcristallin Cellulose; Test type: Superiority or Other; p = 0.25, Fisher Exact
Statistical Analysis 3: Comparison: Saccharomyces Boulardii vs Microcristallin Cellulose; Test type: Superiority or Other; p = 0.87, Log Rank

2. Secondary Outcome: Total Number of Clostridium Difficile-associated Diarrhea Episodes
Time Frame: 29 months
Measure: Number; unit: episodes
Arm/Group | Saccharomyces Boulardii | Microcristallin Cellulose
Number analyzed (Participants) | 246 | 231
episodes | 2 | 2

3. Secondary Outcome: Total Number of Antibiotic-associated Diarrhea Episodes Without Evidence of Clostridium Difficile (Toxins)
Time Frame: 29 months
Measure: Number; unit: episodes
Arm/Group | Saccharomyces Boulardii | Microcristallin Cellulose
Number analyzed (Participants) | 246 | 231
episodes | 19 | 17
Statistical Analysis 1: Comparison: Saccharomyces Boulardii vs Microcristallin Cellulose; Test type: Superiority or Other; p = 0.80, Regression, Cox; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.49 to 1.73]
Statistical Analysis 2: Comparison: Saccharomyces Boulardii vs Microcristallin Cellulose; Test type: Superiority or Other; p = 0.93, Regression, Cox — adjusting for age, sex, CRP, leukocyte count, duration of antibiotic treatment, and administration of antibiotics; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.53 to 2.03]

4. Secondary Outcome: Incidence Density of Antibiotic-associated Diarrhea
Time Frame: 29 months
Measure: Number; unit: cases per year
Arm/Group | Saccharomyces Boulardii | Microcristallin Cellulose
Number analyzed (Participants) | 246 | 231
cases per year | 0.78 | 0.64
Statistical Analysis 1: Comparison: Saccharomyces Boulardii vs Microcristallin Cellulose; Test type: Superiority or Other; p = 0.6, Regression, Logistic — Association between initial leukocyte count and incidence of AAD; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.96 to 1.08]
Statistical Analysis 2: Comparison: Saccharomyces Boulardii vs Microcristallin Cellulose; Test type: Superiority or Other; p = 0.653, Regression, Logistic — Association between the initial C-reactive protein and incidence of AAD; Odds Ratio (OR) = 1.00, 95% CI 2-sided [1.00 to 1.01]

5. Secondary Outcome: Average Duration of Antibiotic-associated Diarrhoea and Clostridium Difficile-associated Diarrhea
Time Frame: 29 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Saccharomyces Boulardii | Microcristallin Cellulose
Number analyzed (Participants) | 246 | 231
days | 4.48 (4.13) | 4.26 (3.85)

6. Secondary Outcome: Average Number of Bowel Movements in Patients With Antibiotic-associated Diarrhoea and Clostridium Difficile-associated Diarrhea
Time Frame: 29 months
Measure: Mean (Standard Deviation); unit: bowel movements per day
Arm/Group | Saccharomyces Boulardii | Microcristallin Cellulose
Number analyzed (Participants) | 246 | 231
bowel movements per day | 4.48 (3.82) | 4.07 (3.13)

7. Secondary Outcome: Total Number of Discontinuation or Change of Initially Prescribed Antibiotic
Time Frame: 29 months
Measure: Number; unit: participants
Arm/Group | Saccharomyces Boulardii | Microcristallin Cellulose
Number analyzed (Participants) | 246 | 231
participants | 14 | 7

ADVERSE EVENTS:
Description: Ten participants did not take trial drug and were excluded from the safety analysis population. Therefore, the numbers of participants at risk are 245 and 222, while the numbers in the participant flow are 246 and 231.
Arm/Group | Saccharomyces Boulardii | Microcristallin Cellulose
Serious Adverse Events (participants affected / at risk) | 9/245 | 3/222
Other Adverse Events (participants affected / at risk) | 9/245 | 9/222
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saccharomyces Boulardii (N=245) | Microcristallin Cellulose (N=222)
Duodenal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Pulmonary empyema (Infections and infestations) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saccharomyces Boulardii (N=245) | Microcristallin Cellulose (N=222)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Faecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Malaise (Gastrointestinal disorders) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No